CLINICAL TRIAL: NCT02170103
Title: Effect of Diagnostic Echocardiogram on Microvascular Recovery Following Acute STEMI
Brief Title: Microvascular Recovery With Ultrasound in Myocardial Infarction (MRUSMI) Post PCI Trial
Acronym: MRUSMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: InCor Heart Institute (Other); VU University of Amsterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0300-17-FB
Record Dates: First submitted 2014-06-13; First posted 2014-06-23 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: STEMI; Chest Pain
Keywords: segment elevation myocardial infarctions (STEMIs),; sonothrombolysis; reperfusion; percutaneous intervention (PCI),; antithrombotic therapy,; antiplatelet therapy,
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Chest Pain | interventions — Percutaneous Coronary Intervention; Microbubbles; perflutren; FS 069; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound and microbubbles (Experimental): Patients who provide emergent consent will be randomized to either conventional therapy for a heart attack, or conventional therapy and ultrasound with microbubbles. The ultrasound will be applied both before and after emergent heart catheterization, in order to break up the blood clots that are not only in the artery supplying the heart muscle, but also in the small branches (capillaries) that are fed by this artery.
  Interventions: Procedure: percutaneous intervention (PCI); Drug: Microbubbles; Procedure: Ultrasound
- Standard of care (Other): Emergent PCI/antithrombotic/antiplatelet therapy with Echocardiogram to assess Left Ventricular Ejection Fraction (LVEF) and Aspirin, Plavix, or Direct Thrombin Inhibitor.
  Interventions: Procedure: percutaneous intervention (PCI)

INTERVENTIONS:
Procedure: percutaneous intervention (PCI) — Successful PCI with the patent vessel and at least Thrombolysis in Myocardial Infarction (TIMI) 2 flow in the left anterior descending artery (LAD) post-PCI.
Drug: Microbubbles — The agents will be divided into two separate doses (two vials per study), and mixed with approximately 29 milliliters of saline (approximately a 2.0-4.0% infusion). The first dilution will be administered pre PCI therapy, and the second dilution infused immediately post PCI. Since Optison is less stable in saline, an alternative approach will be to give the Optison as intermittent 0.1 milliliter boluses followed by 3-5 saline flushes over 10 seconds. The entire duration of each treatment before PCI will be up to 30 minutes depending on time constraints in getting to the catheterization laboratory, while the duration of treatment immediately after PCI will be 30 minutes.
  Other Names: DEFINITY® (Perflutren Lipid Microsphere) manufactured by Lantheus Medical Imaging; OPTISON™ (Perflutren Protein-Type A Microspheres Injectable Suspension, USP) manufactured by General Electric Global Research
  Arms: Ultrasound and microbubbles
Procedure: Ultrasound — Intermittent high Mechanical Index (MI) impulses (0.8-1.4 MI; Frequency 1.0-1.7 MegaHertz (MHz); pulse duration 4-44 microseconds) will be administered over the microvasculature where there are wall motion abnormalities and a perfusion defect using an imaging plane that best aligns itself with the risk area
  Arms: Ultrasound and microbubbles

SUMMARY:
The investigators propose to test the effectiveness of a technique that uses a modified commercially available ultrasound system used for cardiac imaging, and a commercially available ultrasound contrast agent (microbubbles) to break up the blood clots that cause heart attacks. The ultrasound and microbubbles will be applied as soon as possible to patients presenting to the emergency department, after an EKG confirms that a heart attack is ongoing. Patients who provide emergent consent will be randomized to either conventional therapy for a heart attack, or conventional therapy and ultrasound with microbubbles. The ultrasound will be applied both before and after emergent heart catheterization, in order to break up the blood clots that are not only in the artery supplying the heart muscle, but also in the small branches (capillaries) that are fed by this artery. Following the randomized treatment, patients will be followed for the development of any complications (recurrent heart attack, heart failure, or need for defibrillator placement) as well as by echo and cardiac MRI to determine how much heart muscle was salvaged by the treatment.

DETAILED DESCRIPTION:
The investigators propose to test the effectiveness of a technique that uses a modified commercially available ultrasound system used for cardiac imaging, and a commercially available ultrasound contrast agent (microbubbles) to break up the blood clots that cause heart attacks. The ultrasound and microbubbles will be applied as soon as possible to patients presenting to the emergency department, after an EKG confirms that a heart attack is ongoing. Patients who provide emergent consent will be randomized to either conventional therapy for a heart attack, or conventional therapy and ultrasound with microbubbles. The ultrasound will be applied both before and after emergent heart catheterization, in order to break up the blood clots that are not only in the artery supplying the heart muscle, but also in the capillaries that are fed by this artery. Following the randomized treatment, patients will be followed for the development of any complications (recurrent heart attack, heart failure, or need for defibrillator placement) as well as by echo and cardiac MRI to determine how much heart muscle was salvaged by the treatment. A total of 250 patients will be enrolled and followed at two different sites. Randomization will be stratified at each study site. The initial site enrolling patients will be University of Sao Paulo Medical School. The other is Vrije Universiteit (VU) University Medical Center in Amsterdam.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to participating centers with chest pain and EKG evidence of an acute STEMI (two contiguous leads with >0.1 millivolt (mV) ST elevation or >0.1 ST depression in V2-V4) will be asked to participate. The inclusion criteria will be:

  1. Age ≥30 years.
  2. Eligible for emergent PCI/antithrombotic/antiplatelet therapy.
  3. Adequate apical and/or parasternal images by echocardiography.
  4. No contraindications or hypersensitivities to ultrasound contrast agents.

Exclusion Criteria:

1. Known or suspected hypersensitivity to ultrasound contrast agent used for the study.
2. Cardiogenic Shock
3. Life expectancy of less than two months or terminally ill.
4. Known severe cardiomyopathy.
5. Known bleeding diathesis or contraindication to glycoprotein 2b/3a inhibitors, anticoagulants, or aspirin
6. Known large right to left intracardiac shunts.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-16 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
Six month event free survival (EFS) | 6 months
  The time from the start of treatment to first cardiac event or death as a first event. Cardiac events include, congestive heart failure, life threatening arrhythmias, and need for prophylactic defibrillator (primary and secondary).
Myocardial salvageability index | Prior to hospital discharge (48-72 hours)
  The difference between extent of delayed enhancement by Gd MRI and the T2 weighted double or triple inversion spin echo assessment of risk area (defined above).
Frequency of left ventricular remodeling | 6 month follow-up
  Defined as a 20% increase in end diastolic volume at the six month follow up biplane contrast enhanced echocardiogram compared to the pre-discharge contrast enhanced echocardiogram

SECONDARY OUTCOMES:
Safety of contrast in this setting | at the time of procedure to 6 month follow-up
  Assessed by any alterations on oxygen saturation or hemodynamic effects acutely related to ultrasound contrast administration
Frequency of > 50% ST segment resolution by EKG at six hours post PCI. | 6 hours post PCI
  Frequency of > 50% ST segment, (a key indicator for both myocardial ischaemia and necrosis if it goes up or down) resolution by EKG at six hours post PCI.
Area under the Creatine Phosphokinase (CPK) versus time curve | at time of procedure
  Quantifies infarct size
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 120 months
  Defined as the time from the start of randomized treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Porter, MD, Principal Investigator — University of NE Medical Center
Locations (2):
- University of Sao Paulo Medical Center, São Paulo, Brazil
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso JE, Tracy CM, Woo YJ, Zhao DX; CF/AHA Task Force. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2013 Jan 29;127(4):529-55. doi: 10.1161/CIR.0b013e3182742c84. Epub 2012 Dec 17. No abstract available. PMID 23247303
- [Background] Eitel I, Desch S, Fuernau G, Hildebrand L, Gutberlet M, Schuler G, Thiele H. Prognostic significance and determinants of myocardial salvage assessed by cardiovascular magnetic resonance in acute reperfused myocardial infarction. J Am Coll Cardiol. 2010 Jun 1;55(22):2470-9. doi: 10.1016/j.jacc.2010.01.049. PMID 20510214
- [Background] European Heart Rhythm Association; Heart Rhythm Society; Zipes DP, Camm AJ, Borggrefe M, Buxton AE, Chaitman B, Fromer M, Gregoratos G, Klein G, Moss AJ, Myerburg RJ, Priori SG, Quinones MA, Roden DM, Silka MJ, Tracy C, Smith SC Jr, Jacobs AK, Adams CD, Antman EM, Anderson JL, Hunt SA, Halperin JL, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology; American Heart Association Task Force; European Society of Cardiology Committee for Practice Guidelines. ACC/AHA/ESC 2006 guidelines for management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: a report of the American College of Cardiology/American Heart Association Task Force and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Develop Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death). J Am Coll Cardiol. 2006 Sep 5;48(5):e247-346. doi: 10.1016/j.jacc.2006.07.010. No abstract available. PMID 16949478
- [Background] Ross AM, Gibbons RJ, Stone GW, Kloner RA, Alexander RW; AMISTAD-II Investigators. A randomized, double-blinded, placebo-controlled multicenter trial of adenosine as an adjunct to reperfusion in the treatment of acute myocardial infarction (AMISTAD-II). J Am Coll Cardiol. 2005 Jun 7;45(11):1775-80. doi: 10.1016/j.jacc.2005.02.061. PMID 15936605
- [Background] Galiuto L, Garramone B, Scara A, Rebuzzi AG, Crea F, La Torre G, Funaro S, Madonna M, Fedele F, Agati L; AMICI Investigators. The extent of microvascular damage during myocardial contrast echocardiography is superior to other known indexes of post-infarct reperfusion in predicting left ventricular remodeling: results of the multicenter AMICI study. J Am Coll Cardiol. 2008 Feb 5;51(5):552-9. doi: 10.1016/j.jacc.2007.09.051. PMID 18237684
- [Derived] Wu J, Xie F, Lof J, Sayyed S, Porter TR. Utilization of modified diagnostic ultrasound and microbubbles to reduce myocardial infarct size. Heart. 2015 Sep;101(18):1468-74. doi: 10.1136/heartjnl-2015-307625. Epub 2015 Jun 24. PMID 26109588